CLINICAL TRIAL: NCT01884259
Title: Randomised Phase II Pilot Study: Induction Chemotherapy With Docetaxel, Cisplatin and Cetuximab Versus Docetaxel, Cisplatin and 5 FU Followed by Radiotherapy With Cetuximab for Locally Advanced or Not Resectable Carcinoma of the Head and Neck
Brief Title: Induction Chemotherapy With TP+5-FU or TP+Cetuximab Followed by Radioimmuptherapy for Locally Advanced or Not Resectable SCCHNN
Acronym: HNO-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_HNO 2
Record Dates: First submitted 2012-05-18; First posted 2013-06-24 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Squamous Cell Carcinoma of the Hypopharynx Stage III; Squamous Cell Carcinoma of the Hypopharynx Stage IV; Squamous Cell Carcinoma of the Larynx Stage III; Squamous Cell Carcinoma of the Larynx Stage IV; Squamous Cell Carcinoma of the Oropharynx Stage III; Squamous Cell Carcinoma of the Oropharynx Stage IV; Squamous Cell Carcinoma of the Oral Cavity Stage III; Squamous Cell Carcinoma of the Oral Cavity Stage IV
Keywords: local advanced squamous cell carcinoma; Larynx; Hypopharynx; Oropharynx; Cavum oris; docetaxel; cisplatin; 5-fluorouracil; Cetuximab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases | interventions — Docetaxel; Cisplatin; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients receive 3 cycles (cycle duration 21 days) of docetaxel (75mg/m²), cisplatin (75mg/m²) and 5-fluorouracil (750mg/m²) followed by Cetuximab (weekly, starting with 400mg/m² then continuing with 250 mg/m²) with radiotherapy (concomitant boost for 6 weeks).
  Active comparator is 5-fluorouracil for first three cycles.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: 5-fluorouracil; Biological: Cetuximab Radioimmunotherapy; Radiation: Boost irradiation
- B (Experimental): All patients receive 3 cycles (cycle duration 21 days) of docetaxel (75mg/m²), cisplatin (75mg/m²) Cetuximab (weekly, starting with 400mg/m² and continuing with 250 mg/m²), followed by Cetuximab (weekly 250 mg/m²) with radiotherapy (concomitant boost for 6 weeks).
  Experimental: cetuximab for the first three cycles.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Biological: Cetuximab Induction; Biological: Cetuximab Radioimmunotherapy; Radiation: Boost irradiation

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m² on day 1 of 21-days cycle
Drug: Cisplatin — 75 mg/m² on day 1 of 21-days cycle
Drug: 5-fluorouracil — 750 mg/m² day 1 to 5 during 24 hours of 21-days cycle
  Arms: A
Biological: Cetuximab Induction — weekly, starting with 400 mg/m² during 120 min.(saturation) then continuing with 250 mg/m²; duration 3 cycles with 21 days
  Other Names: Erbitux
  Arms: B
Biological: Cetuximab Radioimmunotherapy — weekly, starting with 400 mg/m² during 120 min.(saturation only arm A) then continuing with 250 mg/m²; duration 7 weeks
  Other Names: Erbitux
Radiation: Boost irradiation — First 18 irradiations once daily with single dose of 1,8 Gy for 5 days per week. In addition by day 19 a second irradiation boost will be applied for further 12 days(1,5 Gy per day with at least 5 hours interval to 1,8 Gy dose. This results in total clinical target dose of 72 Gy and total subclinical target dose of 54 Gy. Duration of irradiation: 6 weeks
  Other Names: Concomitant boost-irradiation

SUMMARY:
This multicentre, randomised Phase II Pilot Study evaluates the efficacy of docetaxel, cisplatin and 5-fluorouracil or Cetuximab, followed by Cetuximab with radiotherapy.

DETAILED DESCRIPTION:
It will be evaluated whether 5-FU can be replaced by immunotherapy with cetuximab within a taxane/cisplatin-containing induction-chemotherapy scheme for advanced carcinoma of the head and neck. As 5-FU causes severe mucosal toxicities which are added to known toxicities of cisplatin, a combination-therapy with reduced toxicities and same efficacy would be a acceptable alternative to patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed local advanced squamous cell carcinoma of the Larynx, Hypopharynx, Oropharynx or Cavum oris stage III and IV
* One measureable lesion (CT oder MR)
* Age 18 - 75 (including)
* Performance Score ECOG 0 - 1

Exclusion Criteria selected:

* Distant metastases
* ECOG Score >1
* Prior radiation (Head and neck area)
* Creatinin Clearance below 60 ml/µl
* Acute infections
* Neuropathy grade 3 or 4
* Myocardial Infarction within the last 12 months
* Acute coronary syndrome or othe clinically significant cardiovascular diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2021-01-28 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Response Rate (CR, PR) | 3 months after end of therapy
  RECIST criteria

SECONDARY OUTCOMES:
Overall Response Rate (CR, PR, PD, SD) | until 3 months after therapy
  RECIST
Locoregionally monitoring | after one year
Progression Free Survival (PFS) | 1, 2 and 5 years after start of therapy
Adverse reactions | During treatment and until 60 months after end of radiotherapy
  Information about acute toxicity (grade, relation to study drug) during study treatment and until 3 months after end of radiotherapy will be collected for each patient using CTCAE 3.0 criteria list.
  Information about late toxicity (grade) will be collected after 3 months of radiotherapy and until 60 months after radiotherapy using RTOG/EORTC toxicity criteria.
  Kind and number of toxicities will be described according to grade. The highest grade of each patient and toxicity will be analysed.
Overall-Survival | 1, 2 and 5 years after start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Felix Keil, Prof.Dr., Principal Investigator — Hanuschkrankenhaus
Locations (8):
- Austria (8):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Landesklinikum Krems, Krems
  - Krankenhaus d. Barmherzigen Schwestern Linz, Linz
  - Kepler Universitätsklinikum, Med Campus III. Klinik für Interne 3 - Schwerpunkt Hämatologie u. Onkologie, Linz
  - PMU Salzburg, Salzburg
  - Hanusch Krankenhaus Wien, Vienna
  - Universität f. Strahlentherape, AKH Wien, Vienna
  - Klinikum Kreuzschwestern Wels GmbH, Wels

REFERENCES:
- See also: Sponsor — http://www.agmt.at